CLINICAL TRIAL: NCT04747496
Title: Real-world Study on Edoxaban Treatment in Routine Clinical Practice for Patients With Non-valvular Atrial Fibrillation in China
Brief Title: Real-world Study on Edoxaban Treatment for Patients With Non-valvular Atrial Fibrillation in China
Acronym: ETNA-AF-CHINA
Status: Completed | Type: Observational
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: DSCN-ETNA AF-RWS-001
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Non-valvular Atrial Fibrillation
Keywords: Non-valvular atrial fibrillation; Edoxaban
MeSH Terms: interventions — edoxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- NVAF patients: NVAF adult patients with one or more risk factors treated with edoxaban.
  Interventions: Drug: Edoxaban

INTERVENTIONS:
Drug: Edoxaban — This is a non-interventional, observational study.

SUMMARY:
The safety of edoxaban treatment will be examined using real-world clinical evidence from adult patients with non-valvular atrial fibrillation (NVAF) indications in routine clinical practice.

DETAILED DESCRIPTION:
This non-interventional, observational study will evaluate the safety of edoxaban treatment in adult patients with NVAF indications with one or more risk factors.

The primary objective of the study is to collect and evaluate safety data up to 2 years in a real-world setting in relation to adverse event onset (related to edoxaban treatment), duration, severity, and outcome.

The secondary objective will evaluate the effect of edoxaban treatment on stroke (ischemic and hemorrhagic), systemic embolic event (SEE), transient ischemic attack (TIA), major adverse cardiovascular events (MACE), venous thromboembolism (VTE), acute coronary syndrome (ACS), hospitalization related to cardiovascular condition, extent of exposure and compliance to edoxaban therapy, and rate and reasons of permanent discontinuation of edoxaban therapy.

ELIGIBILITY:
Inclusion Criteria:

* Written, informed consent
* NVAF-patients treated with edoxaban according to packaging information (i.e., for NVAF adult patients with one or more risk factors (such as history of congestive heart failure, hypertension, age ≥75 years old, diabetes, prior stroke or TIA) in prevention of stroke and systemic circulation embolism)
* Not participating in any interventional study at the same time

Exclusion Criteria:

* Not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with NVAF treated with edoxaban will be enrolled in this non-interventional, observational study.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2024-11-27 (Actual)

PRIMARY OUTCOMES:
Incidence (including 95% confidence intervals) of major bleeding events following edoxaban treatment | Baseline up to 2 years post treatment
Incidence (including 95% confidence intervals) of clinically related non-major bleeding events following edoxaban treatment | Baseline up to 2 years post treatment
Incidence (including 95% confidence intervals) of adverse events/adverse drug reactions following edoxaban treatment | Baseline up to 2 years post treatment
Incidence (including 95% confidence intervals) of mortality (cardiovascular and all-cause) following edoxaban treatment | Baseline up to 2 years post treatment

SECONDARY OUTCOMES:
Incidence (including 95% confidence intervals) of stroke (ischemic and hemorrhagic) following edoxaban treatment | Baseline up to 2 years post treatment
Incidence (including 95% confidence intervals) of systemic embolic event (SEE) following edoxaban treatment | Baseline up to 2 years post treatment
Incidence (including 95% confidence intervals) of transient ischemic attack (TIA) following edoxaban treatment | Baseline up to 2 years post treatment
Incidence (including 95% confidence intervals) of major adverse cardiovascular events (MACE) following edoxaban treatment | Baseline up to 2 years post treatment
Incidence (including 95% confidence intervals) of venous thromboembolism (VTE) following edoxaban treatment | Baseline up to 2 years post treatment
Incidence (including 95% confidence intervals) of acute coronary syndrome (ACS) following edoxaban treatment | Baseline up to 2 years post treatment
Incidence (including 95% confidence intervals) of hospitalizations related to cardiovascular condition following edoxaban treatment | Baseline up to 2 years post treatment
Duration of exposure to edoxaban treatment in NVAF patients | Baseline up to 2 years post treatment
Compliance rate of edoxaban treatment in NVAF patients | Baseline up to 2 years post treatment
Proportion of participants who discontinued edoxaban treatment in NVAF patients | Baseline up to 2 years post treatment
Number of interventions related to atrial fibrillation/edoxaban in NVAF patients | Baseline up to 2 years post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (97):
- China (97):
  - Beijing Tsinghua Changgung Hospital Affiliated Hospital of Tsinghua University, Beijing, Changping District
  - Aviation General Hospital of China Medical University, Beijing, Chaoyang District
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Chaoyang District
  - Beijing Chao-Yang Hospital Capital Medical University, Beijing, Chaoyang District
  - Beijing Hospital, Beijing, Dongcheng District
  - Beijing Tongren Hospital,Cmu, Beijing, Dongcheng District
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Guangdong Second Provincial General Hospital, Guangzhou, Guangdong
  - Guangzhou First People'S Hospital, Guangzhou, Guangdong
  - Guangzhou Panyu Central Hospital, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital,Sun Yat-Sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The First People'S Hospital of Nanning, Nanjing, Guangxi
  - The Third People'S Hospital of Nanning, Nanning, Guangxi
  - Heilongjiang Provincial Hospital, Harbin, Heilongjiang
  - Kaifeng Central Hospital, Kaifeng, Henan
  - The Third Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Xinxiang Central Hospital, Xinxiang, Henan
  - The Fifth Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tianjin Medical University General Hospital, Tianjin, Heping District
  - The Second Hospital of Tianjin Medical University, Tianjin, Hexi District
  - Shanghai Ninth People'S Hospital,Shanghai Jiaotong University School of Medicine, Shanghai, Huangpu District
  - Hebei Petro China Center Hospital, Langfang, Hubei
  - Dongfeng General Hospital of Chinese Medicine, Shiyan, Hubei
  - Renmin Hospital of Wuhan University Hubei General Hospital, Wuhan, Hubei
  - The Central Hospital of Wuhan, Wuhan, Hubei
  - Tongji Hospital,Tongji Medical College Huazhong University of Science & Technology, Wuhan, Hubei
  - Union Hospital Affiliated With Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Wuhan Puai Hospital, Wuhan, Hubei
  - Wuhan Third Hospital, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Changsha Central Hospital, Changsha, Hunan
  - Hunan Provincial People'S Hospital, Changsha, Hunan
  - The First Hospital of Changsha, Changsha, Hunan
  - The Fourth Hospital of Changsha, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangtan Central Hospital, Xiangtan, Hunan
  - Changzhou No.2 People'S Hospital, Changzhou, Jiangsu
  - Jiangyin People'S Hospital, Jiangyin, Jiangsu
  - The First People'S Hospital of Kunshan, Kunshan, Jiangsu
  - Jiangxi Provincial People'S Hospital, Nanchang, Jiangsu
  - Nanjing Jiangning Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The Second People'S Hospital of Suzhou, Suzhou, Jiangsu
  - Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu
  - Wuxi People'S Hospital, Wuxi, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Jilin Province People'S Hospital, Changchun, Jilin
  - The Fourth Hospital of Jilin University, Changchun, Jilin
  - The Second Hospital of Jilin University, Changchun, Jilin
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - China Shenyang Chest Hospital, Shenyang, Liaoning
  - The Second Affiliated Hospital of Shenyang Medical College, Shenyang, Liaoning
  - Beijing Miyun District Hospital, Beijing, Minyun District
  - Shanghai East Hospital,Tongji University, Shanghai, Pudong New Area
  - Qingpu Branch of Zhongshan Hospital Affiliated to Fudan University, Shanghai, Qingpu District
  - The Fifth People'S Hospital of Jinan, Jinan, Shandong
  - Affiliated Hospital of Weifang Medical University, Weifang, Shandong
  - Hangzhou Third Hospital, Hangzhou, Shangcheng District
  - Heping Hospital Affiliated to Changzhi Medical College, Changzhi, Shanxi
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Shanxi Cardiovascular Hospital, Taiyuan, Shanxi
  - Shanxi Provincial People'S Hospital, Taiyuan, Shanxi
  - Taiyuan Central Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Beijing Chest Hospital, Capital Medical University, Beijing, Tongzhou District
  - Peking Union Medical College Hospital, Beijing, Xicheng District
  - Peking University First Hospital, Beijing, Xicheng District
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Xuanwu Hospital Capital Medical University, Beijing, Xuanwu District
  - Longhua Hospital Shanghai University of Traditional Chinese Medicine, Shanghai, Xuhui District
  - Shanghai Yangpu East Hospital, Shanghai, Yangpu District
  - The First Hospital of Kunming, Kunming, Yunnan
  - Chongqing General Hospital, Chongqing, Yuzhong District
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Yuzhong District
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Yuzhong District
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Greentown Cardiovascular Hospital, Hangzhou, Zhejiang
  - Zhejiang Hospital, Hangzhou, Zhejiang
  - Zhejiang Provincial Hospital of Chinese Medicine, Hangzhou, Zhejiang
  - Zhejiang Provincial People'S Hospital, Hangzhou, Zhejiang
  - The First Hospital of Jiaxing, Jiaxing, Zhejiang
  - The Second Hospital of Jiaxing, Jiaxing, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Wenzhou Central Hospital, Wenzhou, Zhejiang
  - Wenzhou Hospital of Traditional Chinese Medicine, Wenzhou, Zhejiang
  - Wenzhou People'S Hospital, Wenzhou, Zhejiang
  - Beijing Chao-Yang Hospital Capital Medical University, Beijing
  - Tsinghua University Affiliated Beijing Tsinghua Changgeng Hospital, Beijing
  - The Fourth Hospital of Changhsa, Changsha

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/